CLINICAL TRIAL: NCT03769025
Title: Remote Observed Dosing of Suboxone to Improve Clinical Practice
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kyle Kampman, Medical Director, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RODS; 5U34DA045177-03 (NIH)
Record Dates: First submitted 2018-11-27; First posted 2018-12-07 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Opioid-use Disorder; Opioid Dependence; Opiate Dependence
Keywords: remote observed dosing
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remote Observed Dosing (Experimental): One group will be assigned to Remote Observed Dosing (ROD) and will have all of their Suboxone® doses remotely observed. The intervention is remote observed dosing
  Interventions: Behavioral: Suboxone Remote Observed Dosing
- Attention Control (Active Comparator): The attention control (AC) group will not have their dosing observed but will send a text message confirming they have taken their study medication to the study team daily matching contact with the study team. Text message confirming that they have taken their study medication is the intervention
  Interventions: Other: Suboxone Attention Control

INTERVENTIONS:
Behavioral: Suboxone Remote Observed Dosing — The remote observed dosing group will use the provided smartphone to video record themselves taking their Suboxone dose each day
  Arms: Remote Observed Dosing
Other: Suboxone Attention Control — Attention control group will send a text message daily confirming that they have taken their Suboxone dose
  Arms: Attention Control

SUMMARY:
This is a 15-week, outpatient study of remote observed dosing to improve suboxone compliance in opiate dependent subjects.The main purpose of this study is to see if watching patients take their medication will improve treatment of opiate dependence by prompting patients to take all prescribed doses of Suboxone. Suboxone is approved by the Food and Drug Administration (FDA) for the treatment of opiate dependence. All patients receive a smartphone and patients in the intervention (remote observed dosing) group will use the smartphone to take videos of themselves taking Suboxone.

DETAILED DESCRIPTION:
Opioid use disorder (OUD) is a significant public health problem. About 2 million Americans meet criteria for opioid use disorder involving prescription pain relievers and an additional 591,000 Americans meet criteria for a heroin use disorder. The rise in prescription opioid use in the US has resulted in a dramatic increase in heroin use, as prescription opioid users switch to heroin when their access to prescription opioids become less available. Opioids (including prescription opioids and heroin) killed more than 33,000 people in 2015, more than any year on record. Nearly half of all opioid overdose deaths involve a prescription opioid.

Buprenorphine, a partial agonist that exerts significant actions at the mu opioid receptor, has been shown to be effective for the treatment of OUD. Because it is a partial agonist and not prone to overdose, it is considered to be safe enough to dispense out of a clinician's office as opposed to an opiate treatment program (OTP). The availability of buprenorphine treatment outside of an OTP has significantly expanded the availability of effective treatment for OUD and is associated with reducing disparities related to treatment access.

While initial studies reported little evidence of buprenorphine diversion, more recent studies have indicated buprenorphine is prone to diversion and poor adherence that can significantly diminish its safety and efficacy. In these US clinical trials, adequate adherence to buprenorphine has been shown to occur in fewer than 50% of subjects who are prescribed the medication. In a trial involving 50 African American subjects with opioid use disorder participating in office based buprenorphine treatment, it was found that only 48% of the subjects were adherent to the medication as defined as having 80% or more of their visits associated with a positive UDS for buprenorphine. In another trial involving 703 subjects with opioid use disorder only 41% of the subjects took buprenorphine 80% of the days it was prescribed. Finally in an examination of medical and pharmacy claims data over a year, only 32% of patients participating in office based buprenorphine treatment took buprenorphine on 80% or more days.

Efforts to reduce poor adherence and diversion in buprenorphine maintenance generally include smaller prescriptions and more frequent office visits. An alternative to frequent face to face meetings is using smartphone technology to conduct remote observation of dosing (ROD). In addition, OUD patients have expressed that observed dosing of MMT and flexible dose prescription regimes play an important role in their treatment. However, there have been no published studies using ROD to monitor compliance of Suboxone.

Remote Observed Dosing Intervention We conducted a Stage 1B integrated cellphone based behavioral intervention that visually confirmed medication ingestion, thereby potentially reducing buprenorphine misuse and diversion and improving medication adherence. Patients with OUD, who were not currently prescribed buprenorphine, were recruited. All patients received buprenorphine, a study provided smartphone, weekly Cognitive Behavioral Therapy (CBT), and twice weekly urine screens. The experimental group video recorded themselves taking the medication and these videos were automatically sent daily to the clinical research staff who observed the dosing. This allowed for both the patients and clinical staff to find convenient times to do the tasks and improved clinic office workflow. The attention control (AC) group did not record their medication dosing.

Participants and Recruitment Participants and Eligibility. This study involved individuals with Opioid Use Disorder (OUD) who received three months (12 weeks) of burpenorphine (Suboxone) (standard dose will be up to 16 mgs/day, adjusted as necessary on an individual basis).

Procedures: Patient and Clinical Data Collection Screening Procedures, Suboxone Induction and Randomization. Potential participants will be screened for physical and psychological appropriateness for inclusion in the study using standard intake procedures. Participants who are appropriate for the trial will be inducted onto Suboxone using standard office based induction as described in the ASAM National Practice Guideline for the Use of Medications in the Treatment of Addiction Involving Opioid Use.

Participants will be randomized into one of two study groups based on proportion of use of prescription opiates and heroin, gender, and prior Suboxone treatment. Both groups will receive standard buprenorphine maintenance treatment. Participants will attend study visits twice weekly for 12 weeks. One group will be assigned to Remote Observed Dosing (ROD) and will have all of their Suboxone doses remotely observed using procedures described below. The attention control (AC) group will not have their dosing observed but will send a video message not associated with dosing to the study team daily matching contact time with the study team.

Remote Observed Dosing Compliance. During the start-up phase of the project, we will record a short 5 min instruction video that will be stored on participants' cellphones and on our study web-site that will detail how to take the dosing video and how to ensure it was uploaded correctly. Clinical staff and participants will also be able to use a HIPAA compliant texting service to arrange appointments, send reminders and discuss any study related issues that arise. Note: Participants in the control condition will be provided with a list of prompts and asked to pick one prompt daily to record a video on. They will then follow the same procedures as the experimental condition.

Step 1: Using the study provided smartphone a participant in the experimental condition will use the front facing camera to record taking their study medication.

Step 2: The participant will remove the day's Suboxone dose from their pill pack, place the dose (film) under their tongue and remain with their head in view of the camera until the film dissolves completely. They will then open their mouth, raising their tongue to the roof to ensure the dosage has been dissolved.

Step 3: The participant will end the recording. The phone will automatically save the video onto the micro-sd card and the video will be automatically sent to a secure study server. Once the video is uploaded, a notification message will appear on the participant's phone and the study team will be notified a video has been uploaded. Each recording is expected to last approximately 5 minutes. Note: by saving the video on the micro-sd card, we are safeguarding in the event there is a "bad connection" or "user error" in the video uploading to the server. Phones will be locked with a passcode and if a phone is lost/stolen, it will be "wiped" clean remotely. In addition, a Certificate of Confidentiality will be requested for this research study.

Step 4: Clinical staff will view the video daily. Any instances where the subject moves out of camera view will be recorded as a day without dosing. If the video is not uploaded and is not saved on the micro-sd card, it too will be recorded as a day without dosing.

Step 5: Clinical staff and participants will use a HIPAA compliant text messaging service to communicate. Even though we will train participants on how to take and send dosing videos, we anticipate there will be a slight learning curve. During this time, clinical staff will communicate with participants on how to record the dosing.

All patients who are enrolled will receive a smartphone that includes unlimited talk, text and data. The smartphones will be used to communicate with patients for appointments, make reminder calls, discuss any study related issues, and to record and send the study videos. All patients will be instructed on smartphone use, security and on how to use the phones to record and send the videos to the study team. They will also be instructed about how to take Suboxone and ROD patients will receive additional training on how to ensure the observed dosing video is recorded and uploaded correctly.

Suboxone Dosing. After induction, all patients will receive open-label Suboxone for 12 weeks. Patients in both groups will receive a weeks' worth of Suboxone at each medication management visit. After the 12 weeks of Suboxone, subjects will be referred to on-going treatment options in the community or will be tapered from Suboxone if they so desire.

Cognitive Behavioral Relapse Prevention. In addition to study medication, subjects will participate in weekly, manualized, individual cognitive behavioral relapse prevention psychotherapy. They will also receive weekly Medication Management (MM), adapted for MAT for opioid use disorder.

Weekly visits. Patients will be seen twice weekly. For each in-office visit, patients will provide a urine sample that will be tested for drugs of abuse and for quantitative buprenorphine and norbuprenorphine levels. At each office visit, patients will also complete questionnaires on mood, craving and general health. They will be asked about other medications they are using, about their drug and alcohol use since their last visit, and about any side effects they may be experiencing. Dosage adjustments will be made as needed at the discretion of their clinician.

Medication adherence will be monitored by self-report and verified with creatinine normalized quantitative urinary buprenorphine and norbuprenorphine levels. Urine was chosen as opposed to blood levels to verify adherence for several reasons. First the high number of samples needed to verify adherence over the course of a twelve-week trial would present a great burden to the study patients. Frequent venipunctures can be difficult in patients with opioid use disorder who have a history of IV use of opioids. Creatinine normalized quantitative urine medication levels have been used successfully to verify medication adherence in trials involving both methadone and buprenorphine.

Measures Columbia Suicide Severity Rating Scale (C-SSRS). This is a 5-item scale with additional questions that may be asked based on the participant's responses to the core items. This questionnaire will assess both lifetime and recent suicidal ideation and behavior, including both passive and active thoughts/plans. This data will not be analyzed but will be included to help ensure the safety of the participants.

Timeline Follow Back Interview (TLFB). (The TLFB is a 15-30 minute, semi-structured interview adapted by our laboratory to collect information about daily drug, alcohol, and nicotine use. The TLFB will be given by trained research staff at baseline to cover 3 months immediately preceding treatment entry and will be updated at each research visit to determine any time spent in a controlled environment and cocaine, nicotine, and other drug use during the period since the last visit.

Video Compliance. Submission of videos will be recorded (date and time) and assessed daily for compliance (ie., taking the medication as prescribed). In addition, videos will be saved off the micro-sd cards at each office visit.

Laboratory Measurements (in alphabetical order) Pregnancy Testing. Urine pregnancy tests will be obtained from all women at baseline, week 5, week 9, and end of study.

Quantitative urine buprenorphine and norbuprenorphine levels (using gas chromatography) with urine creatinine used as a control for urinary concentration will be assessed twice weekly throughout the trial. Qualitative (emit) urine toxicology for other drugs (benzodiazepines, barbiturates, opiates, marijuana, methadone, and amphetamine) is done at baseline and weekly throughout the trial.

DATA ANALYSIS For the ROD group, we will calculate the within-patient proportion of study days on which video captured adherence, as per protocol. The primary comparison between the groups will use the creatinine normalized weekly quantitative urine levels for buprenorphine and norbuprenorphine. The main explanatory variable will be a binary indicator for group (ROD vs AC). Our primary analyses will examine the two sets of responses (buprenorphine and norbuprenorphine) separately.

Exploratory Aims Rates of illicit opiate use will be compared between the groups using urine drug screens (UDS) obtained at each visit. A study week will be classified as a "non-use" week if both UDS tests are available and are negative for opiates and if the participant self-reports no use; a study week with a positive UDS or a self-report of use will be classified as a "use" week; study weeks with incomplete data and no test or report of use will be regarded as missing. The number of non-use weeks will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide written informed consent prior to the conduct of any study-related procedure
* Male, female, or transgender
* 18 - 45 years of age
* Meet DSM 5 criteria for opioid use disorder moderate to severe
* Women of childbearing potential must use a reliable means of contraception

Exclusion Criteria:

* Current diagnosis of AIDS
* Participation in buprenorphine maintenance treatment within the past 3 months
* Presence of AST and/or ALT equal to or > 3X upper limit of normal
* Total bilirubin equal to or > 1.5X upper limit of normal and/or estimated creatinine clearance < 60ml/min
* Current diagnosis of pain requiring opioids
* Pregnant or lactating women
* Previous hypersensitivity or allergy to buprenorphine
* Current use of agents metabolized through CYP 3A4 such as azole antifungals (e.g. ketoconazole), macrolide antibiotics (e.g. erythromycin), and protease inhibitors (e.g. ritonavir, indinavir, saquinavir)
* Meet DSM - 5 criteria for current use disorder for any psychoactive substances other than opioids, marijuana, cocaine or nicotine (e.g. alcohol, sedatives)
* Current use of benzodiazepines
* Significant medical or psychiatric symptoms or dementia which in the opinion of the investigators would preclude compliance with the protocol, adequate cooperation in the study, or obtaining informed consent
* Concurrent medical conditions (such as severe respiratory insufficiency) that may prevent the patient from safely participating in the study; and/or any pending legal action that could prohibit participation and/or compliance in study procedures
* Unwilling to accept or use alternative transportation (i.e. public transportation, taxi services, etc.) instead of driving self to appointments during Suboxone Induction
* Living in unstable housing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Kampman, MD, Study Director — University of Pennsylvania; Brenda Curtis, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Treatment Research Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Remote Observed Dosing | Attention Control
Started | 8 | 8
Completed | 3 | 4
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remote Observed Dosing | Attention Control | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (5.1) | 34 (8.4) | 34 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Mean Urinary Buprenorphine Levels
Description: compare the mean urinary buprenorphine level obtained over 12 weeks between the two groups
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Remote Observed Dosing | Attention Control
Number analyzed (Participants) | 8 | 8
ng/ml | 861 (1656) | 287 (253)
Statistical Analysis 1: Comparison: Remote Observed Dosing; Test type: Superiority; p = .1, t-test, 2 sided

2. Secondary Outcome: Percent of Urine Positive Drug Screens
Description: Percent of urine drug screens positive for opiates
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percent of urine positive drug screens
Arm/Group | Remote Observed Dosing | Attention Control
Number analyzed (Participants) | 8 | 8
percent of urine positive drug screens | .3 (.36) | .29 (.49)
Statistical Analysis 1: Comparison: Remote Observed Dosing vs Attention Control; Test type: Superiority; p = .959, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 week
Arm/Group | Remote Observed Dosing | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/8 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remote Observed Dosing (N=8) | Attention Control (N=8)
Diabetic ketoacidosis (Endocrine disorders) | 1 (1) | 0 (0)
nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remote Observed Dosing (N=8) | Attention Control (N=8)
nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
arthralgias (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
fatigue (General disorders) | 1 (1) | 2 (2)
upper respiratory infection (Infections and infestations) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
edema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
drug withdrawal (General disorders) | 2 (2) | 0 (0)
skin infection (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
This trial was intended to be a preliminary trial and involved a small number of subjects. Results should be interpreted accordingly.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT03769025/Prot_SAP_000.pdf